CLINICAL TRIAL: NCT04959890
Title: Methodology Study to Investigate the Utility of Retroviral Insertion Site Analysis in Samples From Subjects Treated With Strimvelis Gene Therapy.
Brief Title: Methodology Study of Retroviral Insertion Site Analysis in Strimvelis Gene Therapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione Telethon (Other)
Responsible Party: Sponsor
Other Study IDs: STRIM-005
Record Dates: First submitted 2021-06-21; First posted 2021-07-13 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Severe Combined Immunodeficiency Due to ADA Deficiency
Keywords: ada-scid; retroviral vector; gene therapy
MeSH Terms: conditions — Severe combined immunodeficiency due to adenosine deaminase deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects Previously Treated with Strimvelis (or GSK2696273) Gene Therapy: It is expected that this study will include approximately 70 eligible samples from approximately 15 subjects previously treated with gamma retroviral gene therapy (gRV-GT).
  Interventions: Genetic: Strimvelis

INTERVENTIONS:
Genetic: Strimvelis — This non-interventional, retrospective, methodology study will use peripheral blood and bone marrow samples previously taken from subjects treated with gRV-GT. The study does not require subjects to undergo any further treatment, intervention or blood withdrawal. Eligible samples will be shipped to a central laboratory and will undergo DNA extraction prior to S-EPTS/LM-PCR analysis. Each analysis run will include a control DNA sample and up to four subject samples. Each sample will be analysed in triplicate.

SUMMARY:
This study is a post approval commitment to evaluate the accuracy and precision of retroviral insertion site (RIS) analysis and its utility for investigating and predicting the potential for insertional oncogenesis in subjects treated with Strimvelis.

DETAILED DESCRIPTION:
This non-interventional, retrospective, methodology study will use peripheral blood and bone marrow samples previously taken from subjects treated with Strimvelis. The study does not require subjects to undergo any further treatment, intervention or blood withdrawal.

The objective of this methodology study is to evaluate the accuracy and precision of shearing extension primer tag selection ligation-mediated polymerase chain reaction (S-EPTS/LM-PCR) for RIS analysis and its utility for investigating and predicting the potential for insertional oncogenesis in subjects previously treated with Strimvelis for severe combined immunodeficiency (SCID) due to adenosine deaminase (ADA) deficiency.

ELIGIBILITY:
Inclusion Criteria

Subjects must have previously received treatment with gRV-GT, either during clinical development (clinical trials and early access programs) or in the post-marketing setting as the approved product (Strimvelis) or under hospital exemption, and for whom at least one biological sample is available that meets the following eligibility criteria::

1. Peripheral blood, bone marrow, or DNA extracted from either source.
2. Taken at least 6 months after gRV-GT.
3. Stored at -20oC or below since the time of sampling.
4. Likely to provide at least 1.5 μg of DNA (following extraction by the central laboratory).

Exclusion Criteria N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will use biological samples previously taken from subjects treated with Strimvelis gRV-GT.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-04-23 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
To assess the precision of S-EPTS/LM-PCR methodology for RIS analysis using control insertion site DNA | Retrospective sample analysis.
  Precision will be determined by the variability (%CV) of the abundance data.
To assess the accuracy of S-EPTS/LM-PCR methodology for RIS using control insertion site DNA | Retrospective sample analysis.
  Accuracy will be determined based on the difference between the mean retrieved abundance and the expected abundance of control DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Fondazione Telethon, Study Director — Fondazione Telethon
Locations (1):
- Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No